CLINICAL TRIAL: NCT06175468
Title: A Randomized, Double-blind, Parallel, Placebo-control Study to Evaluate the Efficacy and Safety of "Formosa 1-Breath Free (NRICM101) " in Subjects With the Symptoms of COVID-19 or Influenza-like
Brief Title: Evaluate the Efficacy and Safety of "Formosa 1-Breath Free (NRICM101) " in Subjects With the Symptoms of COVID-19 or Influenza-like Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: Tian-I Pharmaceutical,. Co. Ltd. (Unknown); China Medical University, China (Other); Qualitix Clinical Research Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMUH112-REC2-154
Record Dates: First submitted 2023-12-13; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Influenza Viral Infections; COVID-19
Keywords: Formosa 1-Breath Free (NRICM101); COVID-19; Influenza
MeSH Terms: conditions — COVID-19; Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo control group (Placebo Comparator): take the placebo drug 5g/bag、three times a day, treatment for 5 days
  Interventions: Drug: Placebo control drug
- Treatment group (Active Comparator): take the Formosa 1-Breath Free (NRICM101) 5g/bag、three times a day, treatment for 5 days
  Interventions: Drug: Formosa 1-Breath Free (NRICM101)

INTERVENTIONS:
Drug: Formosa 1-Breath Free (NRICM101) — After screening, the treatment of this study is divided into two groups: The treatment group is Formosa 1-Breath Free (NRICM101) granule 5g/bag, 3 times a day.
  Arms: Treatment group
Drug: Placebo control drug — After screening, the treatment of this study is divided into two groups: The placebo control group is the placebo (dummy) 5g/bag, 3 times a day.
  Arms: Placebo control group

SUMMARY:
"Formosa 1-Breath Free (NRICM101) " has been widely known in Taiwan to treat COVID-19. However, there is no phase III pivotal clinical trial of "Formosa 1-Breath Free (NRICM101) " . In order to obtain scientific, standardized, and comparable clinical results, the study will be implemented to evaluate the efficacy of safety of "Formosa 1-Breath Free (NRICM101) ".

The objective of the study was used the product which be provided by Tian-I Pharmaceutical Co. Ltd. to evaluate the efficacy and safety of the subjects with the symptoms of COVID-19 or Influenza-like after taking "Formosa 1-Breath Free (NRICM101) ".

This study is a randomized, double-blind, parallel controlled clinical trial. The study consisted of 3 cycles: screening period, treatment period (5 days) and follow-up period. The treatment of this study is divided into two groups: The test drug is Formosa 1-Breath Free (NRICM101) granule 5g/bag, 3 times a day；The control drug is the placebo (dummy) 5g/bag, 3 times a day. The sample size in the study is at least 150 people who can be evaluated, and the dropout rate of the test is 10-15%. The estimated sample size is around 170 people. After signing the ICF, vital signs (sitting blood pressure, pulse rate, SpO2, respiratory rate and body temperature), physical examination, chest X-ray, and laboratory test will be checked in screening period. Only subjects with clinically acceptable and following the inclusion and exclusion criteria will eligible to enroll in this study. Compliance will be assured by administration of the study drug under the supervision of the investigator or his deputy. Subjects will be free to withdraw at any time without stating any reason. Data will be analyzed from those subjects who complete the entire study; however, the case report forms and the final study report should include reasons for withdrawals and any necessary treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet the criteria guideline in the "Seasonal Influenza Prevention and Control Manual" recommended by the Taiwan Centers for Disease Control, or are determined by the investigator to have mild symptoms of COVID-19, including fever, sore throat, cough, and fatigue.
* Subjects who have had a fever (body temperature ≥37.5°C and ≤39°C) before their initial dose.
* Throat pain intensity score >30 points during the screening period.
* Cough severity score >3 points during the screening period.
* Fatigue level score >30 points during the screening period.
* Able to perform activities of daily living and aged 20 weeks or older.
* Duration of illness ≤24 hours.
* Obtained informed consent from the subject and signed the informed consent form.

Exclusion Criteria:

* Subject has used other medications for this condition (including cold medicine, antibiotics, antiviral drugs, and similar traditional Chinese medicines) within the 24 hours prior to screening, or is determined by the investigator to require the use of antibiotics or COVID-19 anti-virus drugs.
* Subject has used corticosteroids or NSAIDs for an extended period within the four weeks prior to screening.
* Subject has had poorly controlled chronic diseases in the past five years, including cardiovascular, respiratory, gastrointestinal, immune-related conditions, or mental health disorders (as determined by the investigator).
* Subject has had chronic bronchitis, streptococcal pharyngitis, herpetic pharyngitis, or pneumonia within the past two years or at the time of screening (as determined by the investigator).
* Subject is allergic to the investigational drug or its components.
* Women who are pregnant, breastfeeding, or planning to become pregnant.
* Subject has participated in other drug clinical trials within the 90 days prior to screening.
* The investigator evaluates the subject unsuitable for inclusion in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Sore Throat Visual Analogue Scale (VAS) | Sore throat will be recorded prior to the first dose, one hour after the first dose every morning, and one hour after the last dose for 5 days
  Assessing the improvement in sore throat in subjects with symptoms of COVID-19 or influenza-like symptoms. Using the Visual Analogue Scale (VAS) with a range of 0-100, the absolute value of the baseline change in pain intensity is calculated as the Sum of Pain Intensity Differences (SPID), serving as an indicator of the degree of therapeutic improvement.

SECONDARY OUTCOMES:
Cough Cough Symptom Score (CSS) | Cough will be recorded prior to the first dose, one hour after the first dose every morning, and one hour after the last dose for 5 days
  Evaluate the improvement in the severity of cough in subjects with symptoms of COVID-19 or influenza-like symptoms. Use the Cough Symptom Score (CSS) to calculate the baseline change as an indicator of the degree of therapeutic improvement.
Fatigue Visual Analogue Scale (VAS) | Fatigue will be recorded prior to the first dose, one hour after the first dose every morning, and one hour after the last dose for 5 days
  Assess the improvement in fatigue in subjects with symptoms of COVID-19 or influenza-like symptoms. Use the Visual Analogue Scale (VAS) with a range of 0-100 as an indicator to calculate the absolute value of baseline change as a measure of therapeutic improvement.
Nasal Symptoms Total Nasal Symptom Score (TNSS) | Nasal symptoms will be recorded prior to the first dose, one hour after the first dose every morning, and one hour after the last dose for 5 days
  Assess the improvement in nasal symptoms in subjects with symptoms of COVID-19 or influenza-like symptoms. Use total nasal symptom score (TNSS) with a range of 0-100 as an indicator to calculate the absolute value of baseline change as a measure of therapeutic improvement.
Fever Level | Fever measurements will be taken before the first dose, and one hour after each dose for 5 days
  Evaluate the improvement in fever in subjects with symptoms of COVID-19 or influenza-like symptoms. Calculate the time (in hours) from the first dose of medication to the first onset of temperature relief, as well as the time from complete relief to a normal value. Temperature relief is defined as a temperature below 37.5°C, and the time for final complete relief is the point in time after the last occurrence of fever when the temperature returns to normal. Additionally, calculate the baseline change in temperature for each measurement as an indicator of therapeutic improvement.
Safety evaluation | Record the adverse event form the baseline to the end of study and follow up to 14 days
  Evaluate the safety of subjects with symptoms of COVID-19 or influenza-like symptoms after administration of the medication to the end of study
Traditional Chinese Medicine (TCM) Syndrome Severity | The Traditional Chinese Medicine (TCM) syndrome will be assessed by the physician during the screening period and at the final follow-up visit up to 14 days.
  Evaluate the improvement in Traditional Chinese Medicine (TCM) syndrome severity in subjects with symptoms of COVID-19 or influenza-like symptoms. Assess the TCM syndrome efficacy using two TCM syndrome scoring scales for primary and secondary symptoms, respectively. Calculate the total scores for the primary symptom scale, the total scores for the secondary symptom scale, and the total syndrome scores (including both primary and secondary symptoms) as indicators of baseline change in absolute values.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ing Li, PhD, Study Chair — Associate Professor
Locations (1):
- China Medical University Hospital, Taichung, Taiwan